CLINICAL TRIAL: NCT06259461
Title: Identifying the Risk of Lung Cancer Linked to Environmental Hormones
Brief Title: Machine Learning to Construct an Association Model for Lung Cancer and Environmental Hormone
Status: Active, not recruiting | Type: Observational
Sponsor: Pei-Hung Liao (Other)
Responsible Party: Sponsor-Investigator, Pei-Hung Liao, Associate Professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Other Study IDs: 202204055RINA
Record Dates: First submitted 2024-01-20; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Lung Neoplasms
Keywords: Environmental Substance
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — (1) 20 years or older; (2) conscious, without mental disorders; (3) able to use Mandarin to communicate, had a smartphone or tablet computer and could operate it by themselves, and were willing to participate in the study after the reasons for participation were explained and a consent form was signed, indicating their consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To apply machine learning to construct an association model regarding lung cancer and environmental hormones to more comprehensively identify factors that may lead to lung cancer and to improve existing lung cancer nursing assessments.

DETAILED DESCRIPTION:
The present study is exploratory, and its design was divided into three stages: Stage 1 explored the environmental hormonal risk factors for lung cancer and constructed an association model using machine learning algorithms. Stage 2 validated the results of the association model with better predictive results in clinical settings. Stage 3 involved recommendations for reconstructing nursing assessments based on the results of the clinical model validation. The three stages are summarized as follows.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years or older;
2. conscious, without mental disorders;
3. able to use Mandarin to communicate, had a smartphone or tablet computer and could operate it by themselves,
4. and were willing to participate in the study after the reasons for participation were explained and a consent form was signed, indicating their consent.

Exclusion Criteria:

* The exclusion criteria were those who could not understand the content of the nursing assessment questions and those with mental disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study focused on lung cancer cases and investigated the association with exposure to environmental hormones
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
identify factors that may lead to lung cancer and environmental hormones. | the database research samples from May 2014 to December 2020.
  This association model can assist in identifying the risk groups of lung cancer and advising physicians on the appropriate environmental hormone testing and treatment to provide nursing guidance and medical advice

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taipei university of nursing and health science, Taipei
  - National Taiwan University, Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: No